CLINICAL TRIAL: NCT04319497
Title: Agreement and Variability of Subjective Refraction, Autorefraction, and Wavefront Aberrometry in Pseudophakic Patients
Brief Title: Subjective and Objective Refraction in Pseudophakic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Refraction
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pseudophakia
Keywords: Subjective Refraction; Autorefraction; Wavefront Aberrometry
MeSH Terms: conditions — Pseudophakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refraction reproducibility and agreement (Other): Subjective and objective refraction will be performed in all patients
  Interventions: Device: Subjective refraction; Device: Autorefraction; Device: Wavefront aberrometry

INTERVENTIONS:
Device: Subjective refraction — Subjective refraction measurements will be performed by two testers for all the patients included
Device: Autorefraction — Five autorefraction measurements will be performed for all the patients included
Device: Wavefront aberrometry — Five wavefront measurements will be performed for all the patients included

SUMMARY:
Targeting of post-cataract refraction depends mainly on the prediction of the post-operative lens position, but also on the post-operative refraction itself. Hence, aim of this study is to evaluate the agreement and variability of subjective refraction performed by two independent examiners, autorefraction, and wavefront aberrometry in pseudophakic patients after uneventful cataract surgery.

DETAILED DESCRIPTION:
One of the main goals of modern cataract surgery, beside removing the cataractous lens, is to achieve the patient's desired post-operative refraction. Targeting this post-operative refraction depends mainly on the prediction of the post-operative lens position and the post-operative refraction itself. Reason for the contributing effect of post-operative refraction in the error-propagation analyses is that refraction in phakic patients was shown to have only moderate reproducibility.

In the past, different studies evaluated refraction methods. However, there is no study that included reproducibility of subjective refraction in pseudophakic patients and compares it with objective refraction methods (autorefraction, wavefront aberrometry).

100 eyes of 100 patients, which underwent uneventful cataract surgery, will be included in the study. Refraction of one eye of each patient will be tested using subjective refraction by two different examiners, autorefraction, and wavefront aberrometry at two separate occasions.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 21 years
* Cataract surgery (at least 8 weeks post-surgery)
* written informed consent

Exclusion Criteria:

* Complications during or after cataract surgery
* Ophthalmic diseases, that might interfere with measurements (macular degeneration, glaucoma, diabetic retinopathia)
* Ophthalmic surgery other than cataract surgery
* Clinically significant posterior capsule opacification

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2014-08-20 (Actual); Study Completion 2014-08-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the agreement between the subjective refraction measurements (in dioptres) of two examiners | 12 months
  To show the number of measurements within the limits of agreement, Bland-Altman plots will be created for subjective refraction measurements in dioptres between examiner 1 and examiner 2.

SECONDARY OUTCOMES:
Evaluation of reproducibility between the subjective refraction measurements between two study visits | 12 months
  To compare reproducibility of subjective refraction measurements between study visit 1 and study visit 2 Wilcoxon-signed rank test will be applied.
Evaluation of the agreement between the measurements performed by subjective refraction, autorefraction, and wavefront aberrometry (in dioptres) | 12 months
  To show the number of measurements within the limits of agreement, Bland-Altman plots will be created for subjective refraction measurements in dioptres between the 3 measurement methods.
Evaluation of the reproducibility between measurements done with subjective refraction, autorefraction, and wavefront aberrometry in dioptres | 12 months
  To compare reproducibility between the 3 measurement methods in dioptres, Friedman's multiple comparison will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Principal Investigator — VIROS, Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiss M, Findl O, Draschl P, Harrer-Seely A, Hirnschall N. Agreement and variability of subjective refraction, autorefraction, and wavefront aberrometry in pseudophakic patients. J Cataract Refract Surg. 2021 Aug 1;47(8):1056-1063. doi: 10.1097/j.jcrs.0000000000000583. PMID 34292891